CLINICAL TRIAL: NCT07106996
Title: Mechanism of Red Yeast Rice Regulating Intestinal Indole Metabolism Pathway to Improve Chronic Inflammation in Polycystic Ovary Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Lishui Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Zhengwei Wan, professor, Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82401924; 8240062474 (Other: the National Natural Science Foundation of China)
Record Dates: First submitted 2025-07-04; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic ovary syndrome; red yeast rice; intestinal microbiota; indole metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accept the red yeast rice intervention group (Experimental): Red yeast rice (RYR), a fermented product that has both medicinal and edible properties, is one of the traditional Chinese medicines used in the treatment of metabolic diseases. The main components of red yeast rice include monacolins, monacolin K, red yeast rice pigments, ergosterol, stigmasterol, β-sitosterol, daucosterol.
  Interventions: Drug: red yeast rice，RYR

INTERVENTIONS:
Drug: red yeast rice，RYR — Participants will take 6 grams of red yeast rice daily for 6 months.

SUMMARY:
The aim of this study is to elucidate the effects of red yeast rice on the improvement of symptoms in patients with polycystic ovary syndrome（PCOS）, and to analyze the dose-response relationship between intestinal microbiota and its metabolite, hydroxyindole, and clinical indicators of PCOS.

The main questions it aims to answer are:

How effective is red yeast rice in treating PCOS? Does the indole metabolic pathway of gut microbiota play a crucial role in the improvement of PCOS symptoms by red yeast rice? Participants will take 6 grams of red yeast rice daily for 6 months, and records will be kept of their PCOS clinical symptoms and indicators before the intervention, at the 3rd month post-intervention, and at the 6th month post-intervention. Additionally, biological samples from feces and serum will be collected at these time points.

ELIGIBILITY:
Inclusion Criteria

* Female patients aged 18-40 years old
* Meeting the Rotterdam criteria (at least two of the following):
* Anovulation or oligo-ovulation
* Clinical evidence of hyperandrogenism or hyperandrogenemia
* Ultrasound findings indicating polycystic ovarian morphology (defined as at least 12 follicles measuring 2-9 mm in diameter and/or an ovarian volume >10 mL [length × width × thickness / 2] in one ovary)
* Subjects who have been fully informed of the study procedures and related risks, and voluntarily agree to participate

Exclusion Criteria

* Pregnant women (confirmed via urine/serum hCG)
* Patients with concomitant infectious diseases or severe dysfunction of multiple systemic organs
* Patients who have taken antibiotics or other drugs (such as probiotics, prebiotics, etc.) that can alter the composition of intestinal flora within 3 months before enrollment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
inflammatory marker IL18 [pg/ml] | Baseline, the 3rd month and the 6th month after the intervention
inflammatory marker IL1β [pg/ml] | Baseline, the 3rd month and the 6th month after the intervention
testosterone (nmol/l) | Baseline, the 3rd month and the 6th month after the intervention
Follicle - Stimulating Hormone (mIU/mL) | Baseline, the 3rd month and the 6th month after the intervention
Luteinizing Hormone (mIU/mL) | Baseline, the 3rd month and the 6th month after the intervention
Estradiol (pmol/l) | Baseline, the 3rd month and the 6th month after the intervention
Progesterone (ng/mL) | Baseline, the 3rd month and the 6th month after the intervention
Prolactin (ng/mL) | Baseline, the 3rd month and the 6th month after the intervention
follicles number | Baseline, the 3rd month and the 6th month after the intervention
  The number of follicles in each ovary of each participant will be determined by ultrasonography.
ovarian volume(Length x Width x Thickness/2,ml) | Baseline, the 3rd month and the 6th month after the intervention
  The size of each ovary in each participant will be determined by ultrasonography.
Follicle diameter(mm) | Baseline, the 3rd month and the 6th month after the intervention
  The diameter of the follicles will be determined by ultrasonography.
Hydroxyindole concentration | Baseline, the 3rd month and the 6th month after the intervention

SECONDARY OUTCOMES:
Body-mass-index (BMI) | Baseline, the 3rd month and the 6th month after the intervention
  BMI measured with the formula BMI=weight [kg]/height² [m]
waist-to-hip ratio | Baseline, the 3rd month and the 6th month after the intervention
  Calculated with the formula: waist circumference/hip circumference

OTHER OUTCOMES:
The metagenomics of fecal samples | before the intervention, at the 3rd month and the 6th month after the intervention
  Total DNA of fecal samples is extracted by CTAB method.
Non-targeted metabolomic analysis of fecal and serum samples | before the intervention, at the 3rd month and the 6th month after the intervention
  Fecal and serum samples were subjected to untargeted metabolomic detection using LC-MS/MS with an Agilent UHPLC system coupled to an Agilent 6538 UHD and Accurate-Mass Q-TOF mass spectrometer. Metabolites in the samples were separated, identified, and their information was acquired. Univariate and multivariate analyses were performed on the metabolites to screen for significantly differential metabolites before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lishui Hospital of Traditional Chinese Medicine, Lishui, Zhejiang, China